CLINICAL TRIAL: NCT04783766
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of CK-3773274 in Healthy Chinese Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics Study of CK-3773274
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: JX01001; CTR20210291 (Other: China CDE clinical trial registration)
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy; Healthy Adult Subjects
Keywords: CK-274; Obstructive hypertrophic cardiomyopathy; CK-3773274; oHCM; aficamten
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- CK-3773274 for Single Ascending Dose (SAD) Cohorts (Experimental): Subjects will be assigned to one of 2 planned dose cohorts and receive single doses of CK-3773274
  Interventions: Drug: CK-3773274
- Placebo comparator for SAD Cohorts (Placebo Comparator): Subjects will be assigned to one of 2 planned dose cohorts and receive single doses of placebo comparator
  Interventions: Drug: Placebo
- CK-3773274 for Multiple Dose (MD) Cohort (Experimental): Subjects will receive multiple doses of CK-3773274
  Interventions: Drug: CK-3773274
- Placebo comparator for MD Cohort (Placebo Comparator): Subjects will receive multiple doses of placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CK-3773274 — CK-3773274- Tablets
  Arms: CK-3773274 for Multiple Dose (MD) Cohort; CK-3773274 for Single Ascending Dose (SAD) Cohorts
Drug: Placebo — Placebo- Tablets
  Arms: Placebo comparator for MD Cohort; Placebo comparator for SAD Cohorts

SUMMARY:
The purposes of this study are to:

1. Learn about the safety of CK-3773274 after a single dose and multiple doses in Chinese healthy adult subjects.
2. Learn how healthy subjects tolerate CK-3773274 after a single dose and multiple doses.
3. Find out how much CK-3773274 is in the blood after a single dose and multiple doses.
4. Determine the effect of doses of CK-3773274 on the pumping function of the heart.
5. Evaluate the effect CYP2D6 genetic polymorphisms on how the body metabolizes CK-3773274.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese males and females between 18 and 45 years of age, inclusive
2. Body weight ≥50kg and body mass index (BMI) within 18 to 26 kg/m2, inclusive
3. Acoustic windows adequate for accurate transthoracic echocardiograms
4. Normal cardiac structure and function, as determined by the cardiologist, or if abnormalities are present, the finding is not clinically significant as determined by the cardiologist
5. LVEF ≥65 percent at screening, and LVEF ≥60 percent at Day-1
6. Normal ECG

Exclusion Criteria:

1. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
2. Subjects with breast implants that may impede echocardiography
3. A clinically significant illness within 4 weeks prior to admission to the CRU
4. Inability to swallow tablets
5. Use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages within 48 hours prior to admission to the CRU
6. Poor peripheral venous access
7. Any blood donation within 60 days prior to admission to the CRU, or any plasma donation within 30 days prior to admission to the CRU, or receipt of blood products within 2 months prior to admission to the CRU

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Subject incidence of Adverse Event (AE), Serious Adverse Event (SAE) | SAD cohorts: Day-1 - Day10; MD cohort: Day-1 - Day 23
Reduced Left Ventricular Ejection Fraction (LVEF) | SAD cohorts: Day-1 - Day10; MD cohort: Day-1 - Day 23

SECONDARY OUTCOMES:
Cmax of CK-3773274 after single and multiple ascending doses | SAD Cohorts: Day-1 - Day10; MD Cohort: Day-1 - Day 23

CONTACTS AND LOCATIONS:
Overall Officials: Chen, MD, Study Director — Corxel Pharmaceuticals
Locations (1):
- Clinical Site, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao X, Liu H, Tian W, Fang L, Yu M, Wu X, Liu A, Wan R, Li L, Luo J, Li Y, Liu B, He Y, Chen X, Li Y, Xu D, Wang H, Han X. Safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of aficamten in healthy Chinese participants: a randomized, double-blind, placebo-controlled, phase 1 study. Front Pharmacol. 2023 Aug 23;14:1227470. doi: 10.3389/fphar.2023.1227470. eCollection 2023. PMID 37680714